CLINICAL TRIAL: NCT05557825
Title: The Use of Photobiomodulation in the Management of Radiotherapy Side Effects: Case Series of Head and Neck Cancer Patients
Brief Title: The Use of Photobiomodulation in the Management of Radiodermatitis in Head and Neck Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Rebeca Boltes Cecatto, Professor Rebeca Boltes Cecatto, University of Nove de Julho
Other Study IDs: Radiodermatite06
Record Dates: First submitted 2022-09-20; First posted 2022-09-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Radiodermatitis; Acute; Radiotherapy Side Effect; Head and Neck Cancer
Keywords: Radiodermatitits; Radiotherapy; Photobiomodulation; Cancer
MeSH Terms: conditions — Radiodermatitis; Radiation Injuries; Head and Neck Neoplasms; Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiodermatitis Case Group: 03 patients with grade 2 to 4 radiodermatitis after radiotherapy for the treatment of head and neck cancer submitted to a PBM/PDT therapy protocol
  Interventions: Radiation: Photobiomodulation Therapy

INTERVENTIONS:
Radiation: Photobiomodulation Therapy — Focal low-level laser therapy, 1 to 3 Joules per point, depending on the degree of pain, wavelength 633 to 830 nm, transcutaneously on the surface of the tissue injured by radiotherapy, three times a week during radiotherapy treatment and two more applications after the end of radiotherapy

SUMMARY:
It is estimated that there will be 670,000 new cases of cancer worldwide in 2020-2022 and it is known that the most commonly instituted treatments in cancer are chemotherapy, radiotherapy and surgery. However, these treatments have undesirable side effects, such as Radiodermatitis after Radiotherapy (RD). In fact, the prevalence of possible side effects after radiotherapy is estimated to be 80 to 90%. Radiotherapy complications are associated with a negative impact on patients' quality of life and few supportive measures are available for such complications. Thus, the management of these side effects has been studied in the literature until the present day. On the other hand, Photobiomodulation (PBM) has an important role in wound repair and tissue regeneration, as it influences the different phases of lesion resolution, including the inflammatory phase, the proliferative phase and the remodeling phase. Thus, the aim of this study is to report a case series of Head and Neck Cancer Patients diagnosed with radiotherapy-induced acute radiodermatitis treated with PBM and/or PDT. This is a case series report and the study data will be extracted from the medical records of threee head and neck cancer patients with grade 2 to 4 followed up from 2022 at the Laser Therapy Outpatient Clinic in a Universitarian Hospital. The outcomes are the size of the lesion, the presence of pain assessed by the Visual Analogue Scale (VAS) and the RTOG Scale (Radiation Therapy Oncology Group Scale) to assess the degree of Radiodermatitis before and after PBM/PDT therapy. Data with positive or negative results will be reported.

DETAILED DESCRIPTION:
It is estimated that there will be 670,000 new cases of cancer worldwide in 2020-2022 and it is known that the most commonly instituted treatments in cancer are chemotherapy, radiotherapy and surgery. However, these treatments have undesirable side effects, such as Radiodermatitis after Radiotherapy (RD). In fact, the prevalence of possible side effects after radiotherapy is estimated to be 80 to 90%. Radiotherapy complications are associated with a negative impact on patients' quality of life and few supportive measures are available for such complications. Thus, the management of these side effects has been studied in the literature until the present day. On the other hand, Photobiomodulation (PBM) has an important role in wound repair and tissue regeneration, as it influences the different phases of lesion resolution, including the inflammatory phase, the proliferative phase and the remodeling phase. Thus, the aim of this study is to report a case series of Head and Neck Cancer Patients diagnosed with radiotherapy-induced acute radiodermatitis Grade 2 to 4, treated with PBM/PDT. This is a case series report and the study data will be extracted from the medical records of three head and neck cancer patients with grade 2 to 4 RD followed up from 2022 at the Laser Therapy Outpatient Clinic in a Universitarian Hospital. The outcomes are the size of the lesion, the presence of pain assessed by the Visual Analogue Scale (VAS) and the RTOG Scale (Radiation Therapy Oncology Group Scale) to assess the degree of Radiodermatitis before and after PBM/PDT therapy. The assessment will be done pre-treatment, weekly during PBM therapy and post-treatment. The PBM therapy are focal low-level laser therapy, 1 to 3 Joules per point, depending on the degree of pain, wavelength 630 to 830 nm, transcutaneously on the surface of the tissue injured by radiotherapy, three times a week during radiotherapy treatment and two more applications after the end of radiotherapy Data with positive or negative results will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of head or neck cancer
* Must be undergoing Radiotherapy
* Must have a diagnosis of Grade II, III or IV radiodermatitis by RTOG Scale, made during the follow-up of the patient in their routine treatment at the hospital by the oncology team
* who do not present clinical signs of another pathology that justifies the presence of the dermis lesion.

Exclusion Criteria:

* Critical clinical states;
* End-of-life or palliative care;
* Patients with skin lesions of another cause even when undergoing RT;
* Patients referred to the laser clinic for the prevention of radiodermatitis without the active RD lesion.
* Patients who have used another photobiomodulation therapy protocol foresaw injury not related to the study.
* All contraindications already defined in the routine referral to the outpatient clinic (patients who have an active tumor at the site to be irradiated; individuals with a history of photosensitivity to photonic or light therapy;patients who have undiagnosed lesions in the treatment region; patients using topical photosensitizing medications or creams;cognitive, psychiatric or neurological changes that prevent the free understanding of the PBM therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: outpatient cancer patients undergoing radiotherapy and who show signs of radiodermatitis RTOG II, III or IV
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Toxicity criteria of the Radiation Therapy Oncology Group Scale (RTOG Scale) | Change from Baseline at 14 days after end of radiotherapy treatment
  RTOG scale assess the degree and intensity of RD. It identifies degree 0 (no reaction), 1 (faint erythema, dry desquamation, epilation, diminished sweating), 2 (moderate, brisk erythema, exudative dermatitis in plaques and moderate edema), 3 (exudative dermatitis, besides cutaneous folds and intense edema) and 4 (ulceration, hemorrhage, necrosis).

SECONDARY OUTCOMES:
Visual Analog Scale of Pain | Change from Baseline at 14 days after end of radiotherapy treatment
  VAS Scale assess the pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

OTHER OUTCOMES:
Lesion Size | Change from Baseline at 14 days after end of radiotherapy treatment
  Evaluation of lesion measurement in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca B Cecatto, M.D. Ph.D., Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho / Post-Graduate program Biophotonics Applied to Health Sciences, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No